CLINICAL TRIAL: NCT00941837
Title: Effect of Dietary Fat Type in Combination With High Protein on Plasma Homocysteine Levels and Selected Markers of Cardiovascular Heart Disease Risk in Human Volunteers
Brief Title: Effect of Dietary Fat Type in Combination With High Protein on Plasma Homocysteine Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Malaysia Palm Oil Board (Other Government)
Collaborators: International Medical University (IMU), Kuala Lumpur,Malaysia (Unknown)
Responsible Party: MPOB, MPOB
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: IMU R043/2008
Record Dates: First submitted 2009-07-16; First posted 2009-07-20 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2011-06

CONDITIONS: Healthy
Keywords: Palm olein; homocsyteine; Cholesterol; lipoproteins; Interleukins; CRP; Blood Pressure; Total homocystein; Serum lipid profile; Serum apolipoproteins; Inflammatory markers
MeSH Terms: interventions — Olive Oil; Coconut Oil

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Olive Oil (Experimental)
  Interventions: Dietary Supplement: Olive Oil, Palm Olein Oil, Coconut Oil
- Coconut oil (Experimental)
  Interventions: Dietary Supplement: Olive Oil, Palm Olein Oil, Coconut Oil
- Palm Olein (Experimental)
  Interventions: Dietary Supplement: Olive Oil, Palm Olein Oil, Coconut Oil

INTERVENTIONS:
Dietary Supplement: Olive Oil, Palm Olein Oil, Coconut Oil — Effect of dietary fat type in combination with high protein on plasma homocysteine levels; 5 wk each with 2 wk wash out in between

SUMMARY:
In this study, the investigators address the research question of whether palm olein will have a positive influence on plasma total homocysteine levels in human volunteers provided with high-protein diets formulated from common Malaysian foods.

Hypothesis: There is a significant difference on the effects of the three experimental oils (palm olein, olive and coconut oil) on plasma tHy levels and the other markers of coronary heart disease (CHD) risk measured.

DETAILED DESCRIPTION:
The experimental are comprise of 30% kcal fat, 20% kcal protein and 50% kcal carbohydrate. Each of the test fat [palm olein (POo), virgin olive oil (OO) and coconut oil (CO)] contributes to two-thirds of total dietary fat will be compared.

Three meals a day providing 2000 kcal, including breakfast, lunch and dinner will be provided for the 5-weeks period of each fat rotation.

45 volunteers are fed with normal cooking oil for 3 weeks for standardisation purpose. They were then stratified into 3 groups according to gender, homocysteine and cholesterol level. The volunteers will be randomized, blinded and will undergo a 3 arms crossover intervention. Each intervention will take 5 wk with 2 wk wash out in between.

Baseline blood samples will be taken while other blood samples will be collected at week-4 and -5 of the study.

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy adult males and females aged 20-60 years, with BMI 23.0 -29.9 kg/m2, and free from any disease (will be decided through history taking, physical examination and biochemical tests).
* Not on any medication or treatment associated with reduction of CHD.
* Non-smokers and non heavy drinker or having smoking or alcoholic history.
* Not pregnant or lactating.
* Willing to adhere to the Dietary Guidelines to the study.

Exclusion Criteria:

* Obese [Body Mass Index (BMI) ≥ 30] or grossly underweight (BMI < 18).
* Suffering from chronic diseases such as diabetes mellitus, CHD, cancer or any liver/renal disease.
* People with blood clotting problem.
* Hypertensive persons (systolic pressure > 140 mmHg, diastolic pressure > 90 mmHg)

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2009-02; Primary Completion 2009-07 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Total homocysteine | 4th and 5th week

SECONDARY OUTCOMES:
Lipids profile and inflammatory markers | 4th and 5th weeks

CONTACTS AND LOCATIONS:
Overall Officials: Voon P T, Principal Investigator — IMU/MPOB
Locations (1):
- Malaysian Palm Oil Board, Kajang, Selangor, Malaysia

REFERENCES:
- [Derived] Voon PT, Ng TK, Lee VK, Nesaretnam K. Virgin olive oil, palm olein and coconut oil diets do not raise cell adhesion molecules and thrombogenicity indices in healthy Malaysian adults. Eur J Clin Nutr. 2015 Jun;69(6):712-6. doi: 10.1038/ejcn.2015.26. Epub 2015 Mar 25. PMID 25804278
- [Derived] Voon PT, Ng TK, Lee VK, Nesaretnam K. Diets high in palmitic acid (16:0), lauric and myristic acids (12:0 + 14:0), or oleic acid (18:1) do not alter postprandial or fasting plasma homocysteine and inflammatory markers in healthy Malaysian adults. Am J Clin Nutr. 2011 Dec;94(6):1451-7. doi: 10.3945/ajcn.111.020107. Epub 2011 Oct 26. PMID 22030224